CLINICAL TRIAL: NCT00988390
Title: Mothers Living With HIV and Their Adolescent Children
Acronym: TALK LA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TALKLA-MH068194; 5R01MH068194 (NIH)
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Family Relations; Mental Health; Physical Health; Risky Sexual Behavior; Substance Use; HIV Infections
Keywords: mothers living with HIV; family intervention; family functioning; conflict; Mental health; and physical health; Family relationships (functioning and conflict)
MeSH Terms: conditions — Psychological Well-Being; Substance-Related Disorders; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention, mothers living with HIV (Other): Mothers living with HIV, Cognitive-behavioral intervention delivered in either English- or Spanish-speaking groups of 5 to 8 mothers living with HIV twice weekly for 1.5 to 2 hours each over eight weeks (n = 16 sessions)
  Interventions: Behavioral: Cognitive-behavioral, small-group format sessions
- Control, mothers living with HIV (No Intervention): Mothers living with HIV, offered intervention at end of study (18 months after recruitment)
- Control, non-HIV-infected mothers (No Intervention): Neighborhood control mothers not infected with HIV, did not receive any intervention

INTERVENTIONS:
Behavioral: Cognitive-behavioral, small-group format sessions — The intervention was delivered in either English- or Spanish-speaking groups of 5 to 8 mothers living with HIV twice weekly for 1.5 to 2 hours each over eight weeks (n = 16 sessions).
  Arms: Intervention, mothers living with HIV

SUMMARY:
* Context: Mothers living with HIV (MLH) and their children face predictable challenges: maintaining physical and mental health, parenting while ill, and addressing HIV-related stressors.
* Objective: To evaluate the efficacy of a family-based intervention over time; to contrast the life adjustments of HIV-affected families and their non-HIV-affected neighbors in the current treatment era.
* Design: Randomized controlled trial of MLH and a longitudinal comparison of MLH to a neighborhood cohort using random effect regression.
* Participants and Intervention: MLH (n = 339) and their school-age children (n = 259) were randomly assigned to receive 1) an intervention of 16 sessions in a cognitive-behavioral, small-group format; or 2) control. MLH and their children were compared to non-HIV-affected families recruited at shopping markets. Participant retention was high: 84% at 6 months, 83% at 12 months, and 78% at 18 months.
* Main Outcome Measures: Family functioning and conflict, mental and physical health, sexual behavior, and substance use.

ELIGIBILITY:
Inclusion Criteria for Intervention/Control, mother living with HIV:

* Mother or primary female caregiver
* Enrolled in HIV-related clinical cares
* At least one child between the age of 6 and 20 years

Inclusion Criteria for neighborhood control, non-HIV-affected mother:

* Mother or primary female caregiver
* not HIV-positive
* At least one child between the age of 6 and 20 years

Exclusion Criteria (Intervention/Control/Neighborhood):

* Mother less than 18 years old
* Unable or willing to give informed consent
* Psychosis or neurological damage as judged by the investigator in consultation with clinical supervisor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2005-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

REFERENCES:
- [Result] Rotheram-Borus MJ, Rice E, Comulada WS, Best K, Elia C, Peters K, Li L, Green S, Valladares E. Intervention outcomes among HIV-affected families over 18 months. AIDS Behav. 2012 Jul;16(5):1265-75. doi: 10.1007/s10461-011-0075-z. PMID 22020758